CLINICAL TRIAL: NCT02630797
Title: Berries and Bones: The Effect of Polyphenolic Metabolites From Blueberries on Bone Turnover
Brief Title: Effect of Blueberries on Bone Turnover
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist - Study Director, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: BB2015
Record Dates: First submitted 2015-12-07; First posted 2015-12-15 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis, Postmenopausal; Bone Loss, Age-related
Keywords: Bone Health; Calcium; Osteoporosis; Polyphenolics
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Intervention Model Description: This partially randomized crossover design model will include participants assigned first to a control baseline period followed by three intervention phases with a low, medium or high daily dose of blueberry products in a randomized order.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Blueberry baseline (Placebo Comparator): No blueberry products provided as part of the usual dietary intake
  Interventions: Dietary Supplement: Blueberry Baseline
- Blueberry Low (Active Comparator): One blueberry product per day containing an equivalent of 0.75 cups of fresh blueberries provided as part of usual dietary intake for 42 days
  Interventions: Dietary Supplement: Blueberry Low
- Blueberry Medium (Active Comparator): Two blueberry products per day containing an equivalent of 1.5 cups of fresh blueberries provided as part of usual dietary intake for 42 days
  Interventions: Dietary Supplement: Blueberry Medium
- Blueberry High (Active Comparator): Four blueberry products per day containing an equivalent of 3 cups of fresh blueberries provided as part of usual dietary intake for 42 days
  Interventions: Dietary Supplement: Blueberry High

INTERVENTIONS:
Dietary Supplement: Blueberry Baseline — Before the study beginning, eligible participants will receive a radioactive tracer, Ca-41, by iv infusion. A total of 150 days will be required for the equilibration of tracer in the body i.e. elimination from soft tissue and deposition in the bone. After equilibration, a baseline period of 42 days will occur, during which no blueberry products will be provided.
  Arms: Blueberry baseline
Dietary Supplement: Blueberry Low — One food or beverage product containing freeze-dried blueberry powder equivalent to 0.75 cups of fresh blueberries will be provided daily for 42 days.
  Arms: Blueberry Low
Dietary Supplement: Blueberry Medium — Two food or beverage products containing freeze-dried blueberry powder equivalent to 1.5 cups of fresh blueberries will be provided daily for 42 days.
  Arms: Blueberry Medium
Dietary Supplement: Blueberry High — Four food or beverage products containing freeze-dried blueberry powder equivalent to 3 cups of fresh blueberries will be provided daily for 42 days.
  Arms: Blueberry High

SUMMARY:
This study uses a bone labeling calcium tracer methodology to compare the dose-response effect of blueberry consumption on calcium retention and bone loss. Post-menopausal women will receive food or beverage products containing freeze-dried blueberries in the amount equivalent to 0.75 (low), 1.5 (medium), and 3 cups (high) of fresh blueberries per day over a 42-day period. The hypothesis is that the polyphenolics found in blueberries will reduce calcium loss from bones.

DETAILED DESCRIPTION:
Participants will be dosed with Ca-41, a rare long-lived radioisotope of calcium. After the equilibration of tracer in the body and its deposition in bones (150 days), subjects will be randomized to one of 6 dose sequences, all of which will begin with a 42-day baseline period. During baseline, 24-hour urine will be collected every 14 days. Following baseline, subjects will enter a 42-day intervention period with one of three doses of blueberries equivalent to 0.75 (low), 1.5 (medium), and 3 cups (high) of blueberries per day. Each dose will be provided in the form of freeze-dried blueberry powder incorporated in 2-4 foods or beverages per day. During the intervention, 24-hour urine will be collected weekly for 6 weeks except week 1. After intervention, subjects will enter a 42-day washout period, during which 24-hour urine will be collected every 3 weeks. The entire study duration will be 444 days for subjects who have not been dosed with Ca-41 previously. In a crossover design, all subjects will complete three 42-day intervention periods corresponding to the three doses of blueberries (low, medium, and high), each followed by a 42-day washout period. The dose-response effect of continuous blueberry consumption over a 42-day period on bone resorption in healthy post-menopausal women will be studied by measuring the loss of Ca-41 in urine by Accelerator Mass Spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Female subject is healthy
* Subject is > 4 years past the onset of natural menopause or total hysterectomy

Exclusion Criteria:

* History of metabolic bone disease or low trauma fractures;
* Subject taking osteoporosis treatment drugs or glucocorticoids within 6 months of the beginning of the study;
* Subjects taking bisphosphonates within 2 years of the beginning of the study;
* History of cancer, thromboembolisms, clotting disorders, uncontrolled hypertension, abnormal thyroid function, malabsorption syndrome, seizure disorders, or heart attack;
* BMI > 35 kg/m2;
* Subjects who will not comply with study interventions ;
* Subjects who will not stop taking natural product supplements of their own selection.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Ca-41 / Ca ratio in 24-hour urinary excretion to estimate calcium loss from bone | From the beginning of baseline (week 0) to the end of the 3rd washout period (week 42)
  Urinary Ca-41 excretion will be expressed as Ca-41/Ca ratio, which is unit-less, and converted to a percent change from the baseline value.
  24-hour urine will be collected approximately every 2 weeks during baseline (week 0, 2, 4, and 6), weekly (except for week 1) during the low, medium, and high blueberry dose interventions completed in a randomized order (weeks 8-12, 20-24, 32-36) and every 3 weeks during the washout periods (weeks 15, 18, 27, 30, 39, 42). Ca-41/Ca ratios will be measured by Accelerator Mass Spectrometry.

SECONDARY OUTCOMES:
Fasting blood and urine analysis of blueberry polyphenolic metabolites | Weeks 0, 6, 12, 18, 24, 30, 36, 42
  Polyphenol concentrations in urine and serum will be expressed in molar units and compared against reference values and across the study periods. Polyphenolic metabolites will be measured by LC-MSMS.
  Fasting blood and urine will be collected at the start and end of baseline (weeks 0 and 6), at the end of the low, medium, and high dose blueberry interventions (weeks 12, 24, and 36), and at the end of the 3 washout periods (weeks 18, 30, 42).
Serum and urine biochemical markers of bone metabolism: calcium concentration | Weeks 0, 6, 12, 18, 24, 30, 36, 42
  Calcium concentration in urine and serum will be expressed in mg/L and measured by Atomic Absorption Spectrophotometry.
  Fasting blood and urine will be collected at the start and end of baseline (weeks 0 and 6), at the end of the low, medium, and high dose blueberry interventions (weeks 12, 24, and 36), and at the end of the 3 washout periods (weeks 18, 30, 42).
Serum biochemical markers of bone metabolism: Insulin Dependent Growth Factor-1 (IGF-1) | Weeks 0, 6, 12, 18, 24, 30, 36, 42
  IGF-1 will be expressed in ng/mL and measured by ELISA.
  Fasting blood will be collected at the start and end of baseline (weeks 0 and 6), at the end of the low, medium, and high dose blueberry interventions (weeks 12, 24, and 36), and at the end of the 3 washout periods (weeks 18, 30, 42).
Serum biochemical markers of bone metabolism: Osteoprotegrin | Weeks 0, 6, 12, 18, 24, 30, 36, 42
  Osteoprotegerin will be expressed in pmol/L and measured by ELISA.
  Fasting blood will be collected at the start and end of baseline (weeks 0 and 6), at the end of the low, medium, and high dose blueberry interventions (weeks 12, 24, and 36), and at the end of the 3 washout periods (weeks 18, 30, 42).
Serum biochemical markers of bone metabolism: RANK ligand | Weeks 0, 6, 12, 18, 24, 30, 36, 42
  RANK-L will be expressed in pmol/L and measured by ELISA.
  Fasting blood will be collected at the start and end of baseline (weeks 0 and 6), at the end of the low, medium, and high dose blueberry interventions (weeks 12, 24, and 36), and at the end of the 3 washout periods (weeks 18, 30, 42).
Serum biochemical markers of bone metabolism: 25(OH) Vitamin D | Weeks 0, 6, 12, 18, 24, 30, 36, 42
  25(OH) Vitamin D will be expressed in ng/mL and measured by LC/MS.
  Fasting blood will be collected at the start and end of baseline (weeks 0 and 6), at the end of the low, medium, and high dose blueberry interventions (weeks 12, 24, and 36), and at the end of the 3 washout periods (weeks 18, 30, 42).
Serum biochemical markers of bone metabolism: Sclerostin | Weeks 0, 6, 12, 18, 24, 30, 36, 42
  Sclerostin will be expressed in ng/mL and measured by ELISA.
  Fasting blood will be collected at the start and end of baseline (weeks 0 and 6), at the end of the low, medium, and high dose blueberry interventions (weeks 12, 24, and 36), and at the end of the 3 washout periods (weeks 18, 30, 42).
Urine biochemical markers of bone metabolism: N-terminal telopeptide (NTX) | Weeks 0, 6, 12, 18, 24, 30, 36, 42
  NTX will be expressed in ng/mL and measured by ELISA.
  Fasting urine will be collected at the start and end of baseline (weeks 0 and 6), at the end of the low, medium, and high dose blueberry interventions (weeks 12, 24, and 36), and at the end of the 3 washout periods (weeks 18, 30, 42).
Serum biochemical markers of bone metabolism: procollagen I intact N-terminal (PINP) | Weeks 0, 6, 12, 18, 24, 30, 36, 42
  PINP will be will be expressed in ug/L and measured by ELISA.
  Fasting blood will be collected at the start and end of baseline (weeks 0 and 6), at the end of the low, medium, and high dose blueberry interventions (weeks 12, 24, and 36), and at the end of the 3 washout periods (weeks 18, 30, 42).

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Weaver, PhD, Principal Investigator — Department of Nutrition Science, Purdue University
Locations (1):
- Department of Nutrition Science Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen JR, Lazarenko OP, Wu X, Kang J, Blackburn ML, Shankar K, Badger TM, Ronis MJ. Dietary-induced serum phenolic acids promote bone growth via p38 MAPK/beta-catenin canonical Wnt signaling. J Bone Miner Res. 2010 Nov;25(11):2399-411. doi: 10.1002/jbmr.137. PMID 20499363
- [Background] Devareddy L, Hooshmand S, Collins JK, Lucas EA, Chai SC, Arjmandi BH. Blueberry prevents bone loss in ovariectomized rat model of postmenopausal osteoporosis. J Nutr Biochem. 2008 Oct;19(10):694-9. doi: 10.1016/j.jnutbio.2007.09.004. Epub 2008 Mar 6. PMID 18328688
- [Background] Weaver CM, Martin BR, Jackson GS, McCabe GP, Nolan JR, McCabe LD, Barnes S, Reinwald S, Boris ME, Peacock M. Antiresorptive effects of phytoestrogen supplements compared with estradiol or risedronate in postmenopausal women using (41)Ca methodology. J Clin Endocrinol Metab. 2009 Oct;94(10):3798-805. doi: 10.1210/jc.2009-0332. Epub 2009 Jul 7. PMID 19584189
- [Derived] Hodges JK, Maiz M, Cao S, Lachcik PJ, Peacock M, McCabe GP, McCabe LD, Cladis DP, Jackson GS, Ferruzzi MG, Lila MA, Bailey RL, Martin BR, Weaver CM. Moderate consumption of freeze-dried blueberry powder increased net bone calcium retention compared with no treatment in healthy postmenopausal women: a randomized crossover trial. Am J Clin Nutr. 2023 Aug;118(2):382-390. doi: 10.1016/j.ajcnut.2023.05.033. Epub 2023 Jun 1. PMID 37269909